CLINICAL TRIAL: NCT06816797
Title: Efficacy of the Cog-Fun Aging Health Promotion Intervention for Older Adults With Subjective Cognitive Decline: A Pilot Controlled Study
Brief Title: Testing the Cog-Fun Aging Program for Older Adults With Subjective Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Principal Investigator, Adina Maeir, Professor Adina Maeir, Hebrew University of Jerusalem
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 20112024
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Subjective Cognitive Decline (SCD); Subjective Cognitive Impairment; Subjective Memory Complaints
Keywords: negative self perceptions; cognitive mistakes; occupational experience; occupational therapy; subjective cognitive decline; health promotion intervention

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from three centers. Each center will form a homogenous group for the Cog-Fun Aging intervention. One center will include both an intervention group and a control group with a crossover component.
  At this center, participants in the intervention group will begin the 10-week Cog-Fun Aging program after an initial baseline assessment (T0). The control group will also be assessed at T0 but will not receive the intervention during this initial phase. Both groups will undergo a second assessment (T1) after the intervention group completes the program to evaluate changes. Following T1, the control group will participate in the intervention and undergo a final assessment (T2) to evaluate the effects of the intervention in the crossover phase. This design allows for comparison between the intervention and control groups, as well as evaluation of outcomes after the crossover phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crossover control group (Experimental): Participants in the control arm will not receive the Cog-Fun Aging intervention during the initial phase (10 weeks). Instead, they will undergo baseline assessments (T0) alongside the intervention group. After the first group completes the 10-week program, the control arm participants will be assessed again (T1). They will then begin the 10-week Cog-Fun Aging intervention and complete a final assessment (T2) after the intervention to evaluate its effects.
  Interventions: Other: Cog-Fun Aging Crossover
- Cog-Fun aging intervention (Experimental)
  Interventions: Other: Cog Fun Ageing intervention

INTERVENTIONS:
Other: Cog Fun Ageing intervention — Cog Fun Aging is a group-based intervention aimed at promoting positive occupational experiences despite cognitive challenges in day to day life. The intervention includes 10 weekly 120-minute group sessions led by experienced occupational therapists. Sessions incorporate learning about the bio-psycho-social factors of SCD and strategies to manage and cope with occupational challenges resulting from SCD.
  Arms: Cog-Fun aging intervention
Other: Cog-Fun Aging Crossover — In the initial phase of the study (between T0 and T1) this group will receive "usual care". Participants are users of regional services where activities for healthy older adults are available. This group will continue going to activities as normal during the initial phase and then participate in the Cog-Fun Aging intervention.
  Arms: Crossover control group

SUMMARY:
The goal of this clinical trial is to learn if the Cog-Fun Aging program helps older adults with Subjective Cognitive Decline (SCD) manage memory challenges and improve their daily lives. The main questions it aims to answer are:

* Does the program help participants better understand their cognitive challenges in daily life?
* Do participants report using more effective strategies to manage their memory difficulties?
* Does the Cog-Fun Aging program reduce negative emotions and self-perceptions related to SCD?

Researchers will compare participants who complete the Cog-Fun Aging program with those who do not to determine the program's effectiveness.

Participants will:

Take part in a 10-week program with weekly sessions. Learn about SCD and how it affects daily life. Practice and monitor strategies to manage memory difficulties.

ELIGIBILITY:
Inclusion Criteria:

* experiencing memory changes and feeling concerned about them
* a score of 23 or higher on the MoCA (Montreal Cognitive Assessment)
* ability to speak and understand Hebrew sufficiently to participate in a Hebrew-speaking group

Exclusion Criteria:

* a self-reported health condition that significantly impacts functioning (e.g., uncontrolled diabetes, severe heart/lung disease)
* residing in a medical institution or nursing home
* currently participating in another SCD treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Memory Impact Questionnaire (MIQ) | After enrollment (before intervention) and 10 weeks later (after intervention)
  The questionnaire was developed for use in both clinical and research settings to better understand the impact of memory changes on the day-to-day functioning of older adults and to monitor outcomes of support programs for this population. In this study the new short form (27 items), not yet published, was used with permission by the authors of the MIQ. The questionnaire includes three subscales: Lifestyle Restrictions (social relationships, work, volunteer and leisure activities), Positive Coping (participation in cognitively engaging tasks and other positive responses to memory changes), and Negative Emotions (negative self-perceptions and perceived negative judgments from others). The total score reflects the overall burden of memory changes, with higher scores indicating with higher scores indicating a greater negative impact. The MIQ has psychometric support, including test-retest reliability (rs = .65-.91) and internal consistency (αs = .87-.93)
Multifactorial Memory Questionnaire-Short Version (MMQ-9) | After enrollment (before intervention) and 10 weeks later (after intervention)
  The short version is a 9 item questionnaire that assesses metamemory. It consists of three scales measuring satisfaction with one's memory (MMQ Satisfaction), self-perception of one's everyday memory abilities (MMQ-Ability), and use of practical memory strategies in day-to-day life (MMQ Strategy). Items are rated on a 5-point Likert scale. The MMQ-9 demonstrates strong psychometric properties, with Cronbach's alpha scores of 0.92 for Satisfaction, 0.86 for Ability, and 0.79 for Strategy, indicating high internal consistency, and intraclass correlation coefficients of 0.89, 0.84, and 0.78, respectively, showing good test-retest reliability. Convergent validity is supported by correlations with related measures (e.g., 0.74 for Satisfaction and 0.70 for Strategy), while discriminant validity is confirmed by negligible correlations with unrelated constructs (e.g., 0.08 for Satisfaction).
Self-Regulation Skills Interview (SRSI) - adpated for study | After enrollment (before intervention) and 10 weeks later (after intervention)
  Evaluates an individual's ability to articulate self-regulation and metacognitive skills in relation to daily life challenges. Includes 6 items that address key domains: emergent awareness, anticipatory awareness, readiness to change, strategy knowledge, strategy use, and strategy effectiveness. In this study, 5 of the 6 items will be utilized, excluding the readiness-to-change domain. Responses are scored on a 10-point scale, and scores are summarized and averaged into two main indices: awareness of difficulties and strategic behavior. Lower scores on these indices indicate stronger abilities in self-monitoring, recognizing, and anticipating difficulties, as well as identifying and effectively applying strategies to manage challenges. The tool demonstrates excellent psychometric properties, with interrater reliability ranging from 0.81 to 0.92 and test-retest reliability between 0.69 and 0.91.
SCD Awareness of Cognitive Difficulties in Daily Life Interview (SCD Interview) | After enrollment (before intervention) and 10 weeks later (after intervention)
  A made-for-study interview to assess participants' ability to describe detailed events in which they encountered cognitive challenges in everyday life and gauge their capacity to identify and articulate the thoughts and emotions that influenced their experiences, the contextual factors that supported or hindered cognitive functioning, the strategies they employed, and how they monitored those strategies' effectiveness in real-time during negative SCD-related daily experiences. Together, the SRSI and the SCD Interview) will provide a comprehensive understanding of participants' awareness of difficulties and strategy use, supporting the evaluation of intervention outcomes.

SECONDARY OUTCOMES:
Patient Health Questionnaire for Depression and Anxiety (PHQ-4) | After enrollment (before intervention) and 10 weeks later (after intervention)
  A 4 item questionnaire that assesses emotional health. The tool combines the PHQ-2 for depression and the GAD-2 for anxiety, featuring a 4-point scale for responses, with total scores ranging from 0 to 12. Higher scores indicate more severe symptoms. The PHQ-4 has strong psychometric support, including internal reliability, construct validity, and factorial validity and criterion validity.

CONTACTS AND LOCATIONS:
Overall Officials: Adina Maeir, PhD, Principal Investigator — School of occupational therapy, faculty of medicine, Hebrew University
Locations (3):
- Israel (3):
  - Hebrew University of Jerusalem, Jerusalem
  - Merhavim Misgav, Misgav Regional Council
  - Hadarim College, Sde Warburg

IPD SHARING:
Plan to Share IPD: No
The study is still in its early stage a research program which aims to enhance the occupational experiences of individuals with Subjective Cognitive Decline (SCD) and identify or develop measures that effectively capture changes in occupational experiences following an intervention. At this stage, the investigators are still assessing whether the data collected by the current measures will adequately reflect the experiences the study seeks to understand and address.

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Ownsworth TL, McFarland KM, Young RM. Development and standardization of the Self-regulation Skills Interview (SRSI): a new clinical assessment tool for acquired brain injury. Clin Neuropsychol. 2000 Feb;14(1):76-92. doi: 10.1076/1385-4046(200002)14:1;1-8;FT076. PMID 10855062
- [Background] Troyer AK, Shaikh KT, Baptist-Mohseni N, Singh A, Duncan-Kofman J, Vandermorris S, Rich JB. Creation and Validation of the MMQ-9: A Short Version of the Multifactorial Memory Questionnaire for Middle-Aged and Older Adults. Clin Gerontol. 2025 May-Jun;48(3):528-538. doi: 10.1080/07317115.2024.2421876. Epub 2024 Oct 29. PMID 39473141
- [Background] Shaikh KT, Tatham EL, Parikh PK, McCreath GA, Rich JB, Troyer AK. Development and Psychometric Validation of a Questionnaire Assessing the Impact of Memory Changes in Older Adults. Gerontologist. 2019 Jul 16;59(4):e248-e257. doi: 10.1093/geront/gny011. PMID 29522122